CLINICAL TRIAL: NCT04274751
Title: Comparison of Transaxillary and Transfemoral Fully-percutaneous Approaches for Transcatheter Aortic Valve Implantation: The TRANSAX Study
Brief Title: Comparison of Transaxillary and Transfemoral Fully-percutaneous Approaches for Transcatheter Aortic Valve Implantation
Acronym: TRANSAX
Status: Completed | Type: Observational
Sponsor: Ignacio J. Amat Santos (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Ignacio J. Amat Santos, Head of Interventional Cardiology Unit, Hospital Clínico Universitario de Valladolid
Organization: Hospital Clínico Universitario de Valladolid (Other)
Other Study IDs: CASVE PI-19-1428
Record Dates: First submitted 2020-01-14; First posted 2020-02-18 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter aortic valve Implantation (TAVI); Transaxillary approach
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transaxillary: TAVI, transaxillary approach
  Interventions: Device: Transcatheter aortic valve implantation
- Transfemoral: TAVI, transfemoral approach
  Interventions: Device: Transcatheter aortic valve implantation

INTERVENTIONS:
Device: Transcatheter aortic valve implantation — Transcatheter aortic valve implantation

SUMMARY:
Retrospective, observational study to compare the outcomes of patient receiving TAVI through transfemoral and transaxillary fully percutaneous approach adjusting for main baseline differences.

DETAILED DESCRIPTION:
Aortic stenosis (AS) is the most frequently treated heart valve disease in our society. Transcatheter aortic valve implantation (TAVI) was originally described through an antegrade transeptal route by Cribier and colleagues in 2002. Because of the complexity of the procedure and risks of damaging the mitral apparatus, this approach was abandoned in favor of less challenging alternatives, with transfemoral (TF) route as primary option. Nevertheless, the TF approach is not feasible or of high risk in between 15 and 35% of the patients and vascular complications have been shown to be an independent predictor of death warranting alternative access techniques for TAVI. In this regard, the transapical, direct aortic, transcarotid, transcaval, and transubclavian/transaxillary (TSc) implantation routes currently serve as alternative access options. The TSc approach was initially used in selected cases. However, recent series suggest that TSc may provide better outcomes than alternative routes when TF is inadequate. Additionally, same studies suggest that, as compared to TF approach, TSc TAVI may present lower rate of vascular complications with comparable rates of other major outcomes despite the worse baseline profile of patients who are considered inappropriate for TF procedures. Moreover, fully-percutaneous TSc approach can be successfully performed with low rate of complications as was recently proposed by some authors. However, comparisons have been based in small series of cases, most of them with former iteration of TAVI devices, and a formal prospective comparison has never been performed. Therefore, our aim is to gather all cases of fully-percutaneous TSc and TF approaches for TAVI in Spain and Portugal and compare the standardized safety and efficacy endpoints through a matched analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent TAVI through transfemoral of transaxillary fully-percutaneous approach between January 2017 and January 2019.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent TAVI through transfemoral of transaxillary fully-percutaneous approach between January 2017 and January 2019.
  All-comers
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
30-day death, stroke or embolic events, PVE or sepsis | 30 day
  Combined endpoint of death, stroke or embolic events, PVE or sepsis at 30-day follow up.
1-year death, stroke or embolic events, PVE or sepsis | 1 year
  Combined endpoint of death, stroke or embolic events, PVE or sepsis at 1-year follow up.
Intraprocedural Vascular complications | Intraprocedural
  Intraprocedural Vascular complications
In-hospital Vascular complications | 7-days
  In-hospital Vascular complications

SECONDARY OUTCOMES:
Short term complications related to the approach. | 30-days
  Short term complications related to the approach.
Mid term complications related to the approach. | 1-year
  Mid term complications related to the approach.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brennan JM, Holmes DR, Sherwood MW, Edwards FH, Carroll JD, Grover FL, Tuzcu EM, Thourani V, Brindis RG, Shahian DM, Svensson LG, O'Brien SM, Shewan CM, Hewitt K, Gammie JS, Rumsfeld JS, Peterson ED, Mack MJ. The association of transcatheter aortic valve replacement availability and hospital aortic valve replacement volume and mortality in the United States. Ann Thorac Surg. 2014 Dec;98(6):2016-22; discussion 2022. doi: 10.1016/j.athoracsur.2014.07.051. Epub 2014 Oct 29. PMID 25443009
- [Background] Cribier A, Eltchaninoff H, Bash A, Borenstein N, Tron C, Bauer F, Derumeaux G, Anselme F, Laborde F, Leon MB. Percutaneous transcatheter implantation of an aortic valve prosthesis for calcific aortic stenosis: first human case description. Circulation. 2002 Dec 10;106(24):3006-8. doi: 10.1161/01.cir.0000047200.36165.b8. PMID 12473543
- [Background] Kurra V, Schoenhagen P, Roselli EE, Kapadia SR, Tuzcu EM, Greenberg R, Akhtar M, Desai MY, Flamm SD, Halliburton SS, Svensson LG, Sola S. Prevalence of significant peripheral artery disease in patients evaluated for percutaneous aortic valve insertion: Preprocedural assessment with multidetector computed tomography. J Thorac Cardiovasc Surg. 2009 May;137(5):1258-64. doi: 10.1016/j.jtcvs.2008.12.013. PMID 19380001
- [Background] Caceres M, Braud R, Roselli EE. The axillary/subclavian artery access route for transcatheter aortic valve replacement: a systematic review of the literature. Ann Thorac Surg. 2012 Mar;93(3):1013-8. doi: 10.1016/j.athoracsur.2011.10.056. Epub 2012 Jan 5. PMID 22226233
- [Background] Walther T, Simon P, Dewey T, Wimmer-Greinecker G, Falk V, Kasimir MT, Doss M, Borger MA, Schuler G, Glogar D, Fehske W, Wolner E, Mohr FW, Mack M. Transapical minimally invasive aortic valve implantation: multicenter experience. Circulation. 2007 Sep 11;116(11 Suppl):I240-5. doi: 10.1161/CIRCULATIONAHA.106.677237. PMID 17846311
- [Background] Bapat V, Khawaja MZ, Attia R, Narayana A, Wilson K, Macgillivray K, Young C, Hancock J, Redwood S, Thomas M. Transaortic Transcatheter Aortic valve implantation using Edwards Sapien valve: a novel approach. Catheter Cardiovasc Interv. 2012 Apr 1;79(5):733-40. doi: 10.1002/ccd.23276. Epub 2011 Sep 26. PMID 21805602
- [Background] Modine T, Sudre A, Delhaye C, Fayad G, Lemesle G, Collet F, Koussa M. Transcutaneous aortic valve implantation using the left carotid access: feasibility and early clinical outcomes. Ann Thorac Surg. 2012 May;93(5):1489-94. doi: 10.1016/j.athoracsur.2012.01.030. Epub 2012 Mar 28. PMID 22464036
- [Background] Greenbaum AB, O'Neill WW, Paone G, Guerrero ME, Wyman JF, Cooper RL, Lederman RJ. Caval-aortic access to allow transcatheter aortic valve replacement in otherwise ineligible patients: initial human experience. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt A):2795-804. doi: 10.1016/j.jacc.2014.04.015. Epub 2014 May 7. PMID 24814495
- [Background] Schofer N, Deuschl F, Conradi L, Lubos E, Schirmer J, Reichenspurner H, Blankenberg S, Treede H, Schafer U. Preferential short cut or alternative route: the transaxillary access for transcatheter aortic valve implantation. J Thorac Dis. 2015 Sep;7(9):1543-7. doi: 10.3978/j.issn.2072-1439.2015.07.27. PMID 26543600
- [Background] Moat NE, Ludman P, de Belder MA, Bridgewater B, Cunningham AD, Young CP, Thomas M, Kovac J, Spyt T, MacCarthy PA, Wendler O, Hildick-Smith D, Davies SW, Trivedi U, Blackman DJ, Levy RD, Brecker SJ, Baumbach A, Daniel T, Gray H, Mullen MJ. Long-term outcomes after transcatheter aortic valve implantation in high-risk patients with severe aortic stenosis: the U.K. TAVI (United Kingdom Transcatheter Aortic Valve Implantation) Registry. J Am Coll Cardiol. 2011 Nov 8;58(20):2130-8. doi: 10.1016/j.jacc.2011.08.050. Epub 2011 Oct 20. PMID 22019110
- [Background] Amat-Santos IJ, Rojas P, Gutierrez H, Vera S, Castrodeza J, Tobar J, Goncalves-Ramirez LR, Carrasco M, Catala P, San Roman JA. Transubclavian approach: A competitive access for transcatheter aortic valve implantation as compared to transfemoral. Catheter Cardiovasc Interv. 2018 Nov 1;92(5):935-944. doi: 10.1002/ccd.27485. Epub 2018 Jan 3. PMID 29314570
- [Background] Garcia DC, Benjo A, Cardoso RN, Macedo FY, Chavez P, Aziz EF, Herzog E, Alam M, de Marchena E. Device stratified comparison among transfemoral, transapical and transubclavian access for Transcatheter Aortic Valve Replacement (TAVR): a meta-analysis. Int J Cardiol. 2014 Mar 15;172(2):e318-21. doi: 10.1016/j.ijcard.2013.12.162. Epub 2014 Jan 9. No abstract available. PMID 24485611
- [Background] Schafer U, Deuschl F, Schofer N, Frerker C, Schmidt T, Kuck KH, Kreidel F, Schirmer J, Mizote I, Reichenspurner H, Blankenberg S, Treede H, Conradi L. Safety and efficacy of the percutaneous transaxillary access for transcatheter aortic valve implantation using various transcatheter heart valves in 100 consecutive patients. Int J Cardiol. 2017 Apr 1;232:247-254. doi: 10.1016/j.ijcard.2017.01.010. Epub 2017 Jan 7. PMID 28118931
- [Result] Amat-Santos IJ, Santos-Martinez S, Conradi L, Taramasso M, Poli A, Romaguera R, Pan M, Bagur R, Del Valle R, Nombela-Franco L, Bhadra OD, Aparisi A, Redondo A, Gutierrez H, Gomez I, Roman JAS. Transaxillary transcatheter ACURATE neo aortic valve implantation - The TRANSAX multicenter study. Catheter Cardiovasc Interv. 2021 Aug 1;98(2):E291-E298. doi: 10.1002/ccd.29423. Epub 2020 Dec 14. PMID 33315296